CLINICAL TRIAL: NCT05002179
Title: Open, Controlled Prospective, Explorative Clinical Trial to Assess Pharmacology and Effectiveness of Echinaforce Chewable Tablets "EC" to Prevent From Enveloped Virus Infections
Brief Title: Echinaforce Study to Investigate Explorative Pharmacology and Effectiveness to Prevent From Enveloped Virus Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Collaborators: CONVEX CRO (Unknown); d.s.h. statistical services GmbH (Unknown); MediStat Ltd. (Unknown); Biodome Clinical (Unknown); Bodimed (Unknown); PPES lab epigenetic signaling (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5'000'760
Record Dates: First submitted 2021-07-08; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Tract Infections; Common Cold
Keywords: SARS-CoV2; Prevention of Respiratory tract infections; Prospective; Controlled; Randomized; Open
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold | interventions — Echinacea extract; Echinaforce

STUDY DESIGN:
Intervention Model Description: Monocentric, 2-armed, randomized, open-label, no-treatment-controlled,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment group, 3 x 2 Echinaforce chewable tablets (EC, 3x800mg) daily during prevention and 5 x 2 EC (5x800mg) during acute viral Respiratory tract infection "vRTIs"
  Interventions: Drug: Echinaforce Chewable tablets
- Control Group (No Intervention): No treatment "Comparison group". Participants are free to take none or any preventive measure. Participants are requested not to take any Echinacea products

INTERVENTIONS:
Drug: Echinaforce Chewable tablets — Preventive treatment: 3X2 EC tablets daily during 2 + 2 months of prevention after run-in of 1 week and intermittent treatment break of 1 week without treatment + 1 month of voluntary follow-up prevention.
  Acute treatment: 5 X 2 EC tablets daily for max. 10 days per individual vRTI or until symptom resolution.
  Other Names: Echinacea; Echinaforce; Echinaforce Junior tablets
  Arms: Treatment group

SUMMARY:
It is a single-center, randomized, open-label, phase IV study for the explorative investigation of the pharmacological mode-of-action of Echinaforce® extract in the form of Echinaforce® Chewable tablets"- Further, it is aimed to evaluate the effectiveness of the study product for the prevention and treatment of respiratory tract infections in generally healthy adults following a real-life setting. The study covers 2x2 + 1 month of prevention in 120 randomized participants following a tight sampling set-up for sensitive detection of viral infections by RT-qPCR analysis of nasal swabs and seroconversion of SARS-CoV2 IgG/IgM in serum samples.

DETAILED DESCRIPTION:
It is a single-center, randomized, open-label, phase IV study for the explorative investigation of the pharmacological mode-of-action of Echinaforce® extract in the form of Echinaforce® Chewable tablets"- Further, it is aimed to evaluate the effectiveness of the study product for the prevention and treatment of respiratory tract infections in generally healthy adults following a real-life setting. The study covers 2x2 + 1 month of prevention in 120 randomized participants following a tight sampling set-up for sensitive detection of viral infections by RT-qPCR analysis of nasal swabs and seroconversion of SARS-CoV2 IgG/IgM in serum samples.

Study flyers are presented in waiting rooms at GPs/hospitals locally and study information is forwarded via the study centre network to attract interest of potential participants. Altogether, 140 participants shall be recruited (screened) by the study. Interested persons shall be invited to the study centre for first informative visit 1 (V1). Participants encountering acute symptoms during screening and/or run-in phase can be included as well. The number of recurrences that can be treated and documented per participant during the time of observation in this study is in principal unlimited. Participants are equipped with study product and study diaries sufficient to encounter a max of 3 individual respiratory tract infections "RTI".

The commercially available study product "Echinaforce Chewable "EC" tablets shall be compared to no treatment in study participants that were randomized equally to the two study groups: 1) "Treatment group" and 2) "no-treatment group". Participants assigned to the "treatment group" are instructed to perform 2 consecutive prevention periods taking 3x2 EC tablets daily for 2x2 months followed by a voluntary, 1 month follow up prevention in frame of this study. After each 2 month prevention phase, participant interrupted prevention for 1 week before starting with a new phase. Intake of regular preventive supplements is recorded as per eCRF entries (V1-V7) and intake of co-medication to treat acute RTI symptoms as per study diary entries. Participants should contact the study coordinator as soon as possible upon first signs of acute cold-/flu like symptoms. The study coordinator confirms the symptoms and instructs participants to start taking 5x2 instead of 3x2 EC tablets daily immediately.

Quality assurance:

Informed Consent Forms, individual e-CRFs accounts and paper study diaries, investigator records, medical test results, and study product must be accessible at all times to study monitors commissioned by the CRO (CONVEX CRO Ltd.) on behalf of and mandated by the sponsor.

The monitor will review the data of the participants and the declared and signed informed consent forms as well as all other study relevant notifications according to procedures defined in the monitoring manual of this study. The monitor will also have access to the source data and undertakes to maintain confidentiality at any time with special regard to reviewed personal, de-anonymized participant data. The monitor assesses protocol deviations of any kind and reports to responsible A. Vogel Clinical trial project manager (CTPM).

In this study, generally, healthy volunteers are to be included and the pharmacological mode-of-action and effectiveness of the test medication, which is Echinaforce Chewable tablets "EC", to prevent from RTIs during phases of prevention assessed with regard to self-diagnosed, usually self-limiting common colds/flu-like infections including infections with SARS-CoV2. Additionally, asymptomatic courses of RTIs are assessed to give a more comprehensive picture of preventive effectiveness. For most of the participants no medical history at the trial center exists and due to the study design, a complete cross-section comparison of e-CRF and participant files waived at the family doctor. With regard to the exclusion criteria (e.g. existence of serious diseases such as autoimmune diseases or degenerative diseases, it is assumed that the participants are aware of them and can name correctly during screening at visit 1). Despite this, no additional comparison between the participant's medical history stored at his doctors place and study centre filed e-CRF accounts/printouts of e-CRF will take place (and vice versa). This also includes relevant AEs/ADRs during the study as well as newly-diagnosed exclusion criteria (accompanying illnesses) during the study period.

The study will be monitored by the executing CRO's representative as specified in the monitoring manual. The monitor will perform an initiation visit before the first participant is screened, have regular contacts with the study site, including routine visits conducted to:

* Provide information and support to the Investigator(s).
* Assure compliance with the study protocol.
* Verify that the research facilities, including laboratories and equipment, are adequate to safely and properly conduct the study.
* Verify that the investigational product is stored properly and under the proper conditions, is in sufficient supply, and that receipt, use, and return of investigational product are controlled and documented adequately.
* Verify that written informed consent was obtained before any protocol-specific screening procedures are performed solely for the purpose of determining eligibility for the clinical study and/or prior to the provision of study product.
* Review the CRFs and source documents to ensure that reported study data are accurate, complete, and verifiable transferred from source documents.
* Ensure that adequate records of clinical trial supplies are maintained.
* Verify that the Investigator and study site personnel are adequately qualified throughout the study.
* Verify that the safety information and amendments are submitted to the relevant authorities and to sponsors.

All checks that the data given in the eCRF complies with the source document will be carried out in accordance with the study specific monitoring manual.

The monitor will be available between visits if the Investigator(s) or other staff at the centre needs information and advice about the study conduct.

After the data base lock and approval from the Sponsor a close-out visit will be performed in order to close the study at the site.

The corresponding SOPs of the executing CRO as well as a study specific monitoring manual set the guidelines applicable for carrying out the monitoring.

The sponsor or a delegate on his behalf, local authorities (Bulgarian drugs administration, BDA) or the responsible ethics committee may inspect this study to reassure quality. The inspectors must be granted access to all medical documents, study documents, correspondence and declarations of consent of participants, which are deemed relevant. All parties involved are to uphold the confidentiality regarding all de-anonymized participant data.

Source data/SDV:

Source data are the original records of all variables collected for the clinical investigation. They include:

* Signed informed consent
* Original printouts of laboratory reports.
* Progress notes, Follow-up notes.
* All filled-out S/AE forms.
* Filled study diaries.
* Descriptions of interventions done to the participants in the study.
* Original Data Records kept at the pharmacy, laboratory or any other 3rd party vendor involved in this study
* Evaluation checklists
* Study product related records (dispensation, return, replacement, compliance, etc.).
* Documentation of sample storage, processing and shipment. The Investigator must allow the monitor access to all documents in the participant's study file to confirm their consistency with the eCRF entries. All study data will be handled confidentially. No information about participant identity on these documents will be allowed to leave the study site.

It is the responsibility of the Investigator to maintain a comprehensive and centralized filing system of all relevant documentation.

• Investigators will be instructed to retain all study records required by the Sponsor and regulatory authorities in a secure and safe facility with limited access for one of the following time periods based on notification from the Sponsor:

* For a period of at least 2 years from the last marketing approval worldwide or for at least 25 years, whichever is the greater
* Or a period of at least two years after discontinuation of clinical development of the investigational product as confirmed by the Sponsor
* For a longer period if required by local regulations The Investigator will be instructed to consult with the Sponsor before disposal of any study records and to provide written notification to the Sponsor of any change in the location, disposition, or custody of the study files.

The sponsor or its representative may visit the study facilities at any time in order to maintain current and personal knowledge of the study through review of the records, comparison with source documents, observation and discussion of the conduct and progress of the study. The investigator will permit trial-related monitoring, audits, EC review and regulatory inspections, providing direct access to source data and study documents

Data coding:

The full details of procedures for data handling will be documented in the Data Management Plan (DMP).

AEs and medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 17.1GE). Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary.

Unique numbers will identify the participant and the biological material obtained from the participant. Appropriate measures such as encryption or deletion will be enforced to protect the identity of human participants in all presentations and publications as required by local/regional/national requirements.

Sample size assessment:

A sample size calculation has been conducted on the main study parameter, which is the incidence of RTIs during the time of observation. A difference between both study groups of at least 20.5% will be recognized as significant clinically relevant (two-group Chi-square test with a 0.05 two sided significance level) with a power of 80% with an incidence rate of 10% seen under active treatment and at least 60 participants included evaluable per study group (chi²-test, nquery advisor 7.0). In addition, for the pharmacological parameters assessed in the study it is estimated that 80% power is achieved with cross-sectional and longitudinal sampling to detect CpG DNA methylation differences of 20%.Amendments to the protocol

SAP:

For planning the statistical analysis and reporting in this clinical study the ICH guidelines for "biostatistical methodology in clinical trials" are taken into account. The details of the statistical methodology (including the handling of missing and incorrect data) are presented in detail in a separate statistical analysis plan (SAP).

Descriptive parameters are determined for assessed clinical variables. In addition to the absolute and relative frequencies of the score values, the arithmetic mean, median, first and third quartile (Q1 or Q3), standard deviation, minimum and maximum of the current value and the changes in comparison between "treatment group" and "no treatment group", are calculated. All assessed target variables are exploratory evaluated using suitable test methods (Mantel-Haenszel test for ordinal variables, Fisher's exact/Chi-Square test for dichotomous or categorical variables and t-test or analysis of variance for quantitative target variables) in the "treatment group" compared to "no treatment group".

The safety assessment is based on the recording of adverse events (AEs), adverse drug reactions (ADRs) as per entries in the e-CRF and ultimately the subjective assessment of tolerability and acceptance by the study investigators and participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years.
* Written informed consent.
* Good knowledge of respective language.
* Willingness to give swab samples.
* Willingness to give blood and saliva samples.

Exclusion Criteria:

* ≥76 years
* < 18 years.
* Participation in another clinical study in the past 30 days or planned during study conduct.
* Permanent intake of antimicrobial, antiviral, immune suppressive substances.
* Surgical intervention in the 3 months prior enrolment or planned intervention during the study conduct.
* Known diabetes mellitus.
* Known atopy (a constitution to produce an exaggerated immune response to otherwise harmless environmental substances, with clinical manifestation of an allergic disease such as allergic rhinitis, eczema, asthma, atopic dermatitis, etc.)
* Cystic Fibrosis, bronchopulmonary dysfunction, COPD.
* Known immune system disorders and degenerative disorders (autoimmune disorders, AIDS, leukaemia, lymphoma, myeloma).
* Known metabolic or resorption disorders.
* Known liver or kidney illnesses (chronic hepatitis, liver cirrhosis, chronic kidney insufficiency).
* Serious health conditions (limited general condition, auto-immune diseases, tumorous diseases, neurological disorders)
* Known allergies to plants of the compositae family (e.g. camomile or dandelion) or one of the compounds in the investigational product
* Known or planned pregnancy during study period (effective contraception is required).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory tract infections "vRTIs" with treatment in comparison to no treatment | 5 months
  The incidence of respiratory tract infections "vRTIs" with treatment in comparison to no treatment is determined as per study diary entries (acute symptomatic episodes of RTIs), by taking nasal swab samples and blood samples from participants during prevention and acute vRTIs. Swab samples are taken by using validated swab sticks (COPAN) and presence of viral RNA/DNA determined by using the RT-PCR respiratory pathogen panel from VIASURE ®, plus a separate panel for SARS-CoV2. Seroconversion of SARS-CoV2 specific IgG/IgM levels is used to detect additional asymptomatic vRTIs. Analyses are done by a non-parametric Chi-square test

SECONDARY OUTCOMES:
Changes of viral load and incidence of responder | 5 months
  The number of participants per time point that become RT-PCR negative is deduced from RT-PCR by means of absolute and relative changes of viral load as per Ct values is determined. Swab samples are taken from participants during prevention and acute vRTIs. Swab samples are taken by using validated swab sticks (COPAN) and presence of viral RNA/DNA determined by using the RT-PCR respiratory pathogen panel from VIASURE ®, plus a separate panel for SARS-CoV2
Development of symptom scores of respiratory tract infections | 5 months
  Development of symptom courses and Total symptom score "TSSc" of all symptoms as per study diary entries. Cold symptoms that are assessed: Runny nose, Congested nose, Sneezing, Cough, Shivering, Malaise, Fatigue/Tiredness, Headache, Myalgia, Anosmia, Insomnia, Sore throat, as Total sum symptom score "TSSc" and individual symptom courses (Scale: absent=0 to severe = 3). Cold symptoms are rated individually for each individual vRTI and the sum score of all rated symptoms together per time point depicts the total symptom score "TSSc". The body temperature is determined in °C by means of an electronic thermometer. The analysis is done by parametric (ANOVA) and non-parametric (chi-square, logistic regression) endpoint analysis
Duration of respiratory tract infections | 5 months
  The duration of vRTIs is determined by Kaplan-Meier analysis until TSSc or individual symptoms scores reach a final score of 1/0 and body temperature reaches <38 °C. The analysis is done by parametric (ANOVA) and non-parametric (chi-square, logistic regression) endpoint analysis
Incidence rate of respiratory tract infections complications, recurrences and antibiotic use | 5 months
  The rate of complications (pneumonia, bronchitis, sinusitis), recurrences and antibiotic use during vRTIs is assessed as per study diary and eCRF entries. Rate and kind of complications and antibiotic use are assessed. The analysis is done by non-parametric Chi-square test
Cumulative number of sick days | 5 months
  The number of sick days during the time of observation in this study is assessed as per study diary entries. A sick day is defined as: day with minimum 1 symptom of a minimally mild symptom severity score of > 0). The analysis is done by non-parametric Chi-square test.
Rate of lost work and lost school days. | 5 months
  The rate of lost work and school days during acute vRTIs is assessed as per study diary and eCRF entries. The analysis is done by non-parametric Chi-square test.
Incidence of household members of participants with acute cold/flu symptoms and confirmed SARS-CoV2/Influenza infections. | 5 months
  The incidence rate of participants' household member with acute cold/flu-like symptoms and/or confirmed SARS-CoV2/Influenza infections is assessed as per eCRF entries by asking participants regularly upon study centre visits. The analysis is done by non-parametric Chi-square test.
Explorative assessment of the absolute and relative changes in the concentration of immunoglobulin-levels (IgM/IgG) | 5 months
  The pharmacological mode-of-action of Echinaforce® extract is investigated by determining absolute and relative changes of immunoglobulin-levels (IgM/IgG) relative to baseline in cross-comparison between study groups and biological samples, (ie. Swab, blood and saliva) from participants with or without (viral)RTIs. The analysis is done by parametric (ANOVA) and non-parametric (chi-square, logistic regression) endpoint analysis
Explorative assessment of the absolute and relative changes in the concentration of cytokine/chemokine-levels | 5 months
  The pharmacological mode-of-action of Echinaforce® extract is investigated by determining absolute and relative changes of cytokine/chemokines-levels analyzed by ELISA analyses relative to baseline in cross-comparison between study groups and biological samples, (ie. Swab, blood and saliva) from participants with or without (viral)RTIs. The analysis is done by parametric (ANOVA) and non-parametric (chi-square, logistic regression) endpoint analysis
Explorative assessment of the absolute and relative changes of the Degree of epigenetic modifications | 5 months
  The pharmacological mode-of-action of Echinaforce® extract is investigated by determining absolute and relative changes of the degree of epigenetic modification analyzed by immunomethylomics assays relative to baseline and in cross-comparison between study groups and biological samples, (ie. Swab, blood and saliva) from participants with or without (viral)RTIs. The analysis is done by parametric (ANOVA) and non-parametric (chi-square, logistic regression) endpoint Analysis.
Change of subjective impression of resistance status during the time of observation | 5 months
  The change of the individual resistance status and resistance against infectious diseases during the time of observation in this study is assessed by asking the participant upon inclusion visit 1 (V1) and at the end of the study upon final visit 6 (V6): how she/he would assess his/her immune status and/or its change under treatment in comparison to assessment during run-in week?) on a scale: bad = 0, average = 1, good = 2, very good = 3.)
Absolute and relative change of sleep quality | 5 months
  The sleep quality are assessed as per eCRF entries by filling the validated Pittsburgh Sleep Quality index (PSQI) at inclusion visit (V1) and final visit 6 (V6) by the participant. The scores are calculated according to validated procedures and the absolute scores and relative changes during the course of the study at the end of prevention (V6) in comparison to baseline (V1) determined
Absolute and relative change of perceived stress. | 5 months
  The perceived stress is assessed as per eCRF entries by filling the validated Perceived Stress Score index (PSS) at inclusion visit (V1) and final visit 6 (V6) by the participant. The score is calculated according to validated procedures and the absolute scores and relative changes during the course of the study at the end of prevention (V6) in comparison to baseline (V1) determined
Subjective treatment effectiveness in view of participants | 5 months
  The subjective treatment effectiveness is rated by the participants of the treatment group at the end of prevention upon final visit (V6) as per eCRF entries by asking the question how the participant would rate the effectiveness of EC tablets to prevent from vRTI pathologies. by asking how effective EC tablets apparently reduced duration and severity of vRTI symptoms?) on a scale: bad = 0, average = 1, good = 2, very good = 3. Rating effectiveness is "n/a = not applicable" for participants assigned to the no treatment group]
Subjective treatment effectiveness in view of investigator | 5 months
  The subjective treatment effectiveness is rated by the investigator for participants of the treatment group at the end of acute vRTIs (VA4) as per study diary entries and eCRF entries (study investigator) by asking the investigator, how effective EC tablets apparently reduced duration and severity of vRTI symptoms in participants treated?) on a scale: bad = 0, average = 1, good = 2, very good = 3. Rating effectiveness is "n/a = not applicable" for participants assigned to the no treatment group]
Incidence and severity of symptoms other than those recorded in the study diary (S/AE) | 5 months
  [(S)AE, occurring during the conduct of this study are detected as per e-CRF entries upon study centre visits (by asking participants of both study groups the question whether any abnormal incidents/symptoms next to cold/flu symptoms occurred during treatment?). Such events are additionally assessed after termination of the study in the form of a compiled safety report
Assessment of subjective rating of tolerability | 5 months
  The treatment tolerability is assessed by participants of the treatment group and the study investigator at the end of prevention upon final visit (V6) as per eCRF entries by asking the question how they rate the tolerability of EC tablets on a scale: bad = 0, average = 1, good = 2, very good = 3). Participants assigned to the no treatment group omit rating the tolerability
Preventive supplements, concomitant medication and -therapies. | 5 months
  The use of any regular preventive supplements in addition to EC tablets is assessed as per eCRF entries. Participants of both study groups are asked about the use of any such product during the time since last visit frequently during study centre visits. By asking if they have taken any preventive supplement regularly during the past month (at least every 2nd day or 2 weeks of the past month)?. The use concomitant medication/therapies for the treatment of acute symptoms of vRTI including antibiotics is assessed as per study diary entries and by asking participants upon study centre visits VA1, VA2, VA3, VA4 the question whether they took any medication/therapy to treat symptoms of vRTIs and if yes, which ones (full product name, dosing, duration) and to treat which symptoms?. The analysis is done by non-parametric chi-square endpoint analysis]
Assesment of subjective ratings of acceptance | 5 months
  The acceptance of the preventive treatment by participants of the treatment group is assessed by e-CRF entries at the end of prevention (V6) (by asking the question whether or not the participant would retake the take EC tablets again for the prevention of vRTIs complaints?). Participants assigned to the no treatment group omit assessing the acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kolev, Dr. med., Principal Investigator — Diagnostics and Consultation Center Convex
Locations (1):
- Diagnostics and Consultation Center Convex EOOD, Sofia, Bulgaria